CLINICAL TRIAL: NCT06634134
Title: Hoe Fietst de Vrouwelijke Wielrenner Door Haar Menstruatiecyclus?
Brief Title: Cycling Through the Menstrual Cycle
Status: Recruiting | Type: Observational
Sponsor: Martini Hospital Groningen (Other)
Collaborators: Antonius Ziekenhuis (Unknown); Reinier de Graaf Groep (Other); sportgeneeskunde Friesland (Unknown); sport medisch centrum tilburg (Unknown)
Responsible Party: Sponsor
Other Study IDs: MenstrualCycling
Record Dates: First submitted 2024-08-15; First posted 2024-10-09 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Menstrual Cycle-based Periodized Training; Female Athlete Triad; Menstrual Cycle
Keywords: Menstrual Cycle; Artificial Intelligence; Cycling; Female Athlete Triad; Female Athletes; Menstrual Cycle-based Periodized training
MeSH Terms: conditions — Female Athlete Triad Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female cyclist: All female cyclist that consent using the data collected by JOIN cycling app and also give permission tracking thier menstrual cycle.
  Natrual menstrual cycle. Hormonal contraceptive use Intra-uterine device use (hormonal vs non-hormonal)
  Interventions: Behavioral: Adjusting training advice

INTERVENTIONS:
Behavioral: Adjusting training advice — Based on discomfort related to the menstrual cycle the female cyclist can choose to adjust the suggested training.

SUMMARY:
With an increase in number of female athletes in sport events, it is becoming more important to gain insight in female related sports physiology. A main difference between male anf female athletes is the menstrual cycle. During the menstrual cycle, female reproductive hormones fluctuate. These hormones are also of influence on endurance, recovery, muscle strenght and mental state. Therefore we hypothesize that training efficiancy, power and motivation to train differ during the menstrual cycle. In case there is a pattern seen during the menstrual cycle, training programs can be individualized taking the menstrual cycle into account leading to more effective training programs.

DETAILED DESCRIPTION:
More and more women are trying to take their menstrual cycle into account when it comes to training effort, planning and performance. This is called menstrual cycle-based periodized training. However, it is still unknown what the exact influence of the different phases of the menstrual cycle is on training and performance. This includes the influence of hormonal fluctuations during the cycle on training capacity, effort load, restorative capacity, motivation to train and perform, daring to take risks and the mental aspects surrounding training and performance. As a result, general advice about cycle-based periodized training cannot be given at this time.

It has been described in the literature that professional-level cyclists regularly have menstrual cycle disorders (ie RED-s). This has short-term health consequences (less rapid recovery, fatigue) and long-term (osteoporosis, increased risk of cardiovascular disease). At a professional level, this knowledge is slowly penetrating. Less is known about the menstrual cycle of amateur athletes and there is also a lack of knowledge about the effects of the menstrual cycle on performance (endurance capacity, heart rate zones, power achieved).

To gain more insight into the menstrual cycle, the influence of the cycle on training and performance and the influence of training on the cycle of the sporting woman, the aim of this study is to monitor the menstrual cycle of female cyclists in combination with their subjective and objective training parameters. This allows us to create insight and, if useful, adapt training on an individual basis to the phase of the menstrual cycle.

The aim of this research is to investigate how the cyclists' menstrual cycle progresses and whether the cycle has an effect on performance.

ELIGIBILITY:
Inclusion Criteria:

* JOIN cycling app member
* female cyclist
* informed consent period tracking in JOIN

Exclusion Criteria:

* none

Ages: 12 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Female JOIN cycling app members that consent with tracking the menstrual cycle.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Health of menstrual cycle in amateur cyclist | 1 year
  It is known that the incidence of amenorrhea is about 15% of the professional female athletes. This has many short- and long term health consequences. These health consequences can be avoided since developing amenorrhea is preventable. It is unknown how many amateur cyclist have an irregular period or have amenorrhea. Insight in the size of this health problem creates a window of opportunity in preventive medicine.
Objective training parameters during the menstral cycle | 2 years
  By collecting details in regards to the menstrual cycle in combination with objective parameters (heart rate, power, speed, endurance) of training it is possible to investigate whether these objective parameters are influenced by the hormonal fluctuations during the menstrual cycle.
Subjective training parameters during the menstrual cycle | 2 years
  By collecting details in regards to the menstrual cycle in combination with subjective parameters (fatigue, discomfort, readiness, motivation) of training it is possible to investigate whether these subjective parameters are influenced by the hormonal fluctuations during the menstrual cycle.

SECONDARY OUTCOMES:
Is menstrual cycle-based periodized training feasible in the future? | 2 years
  In case the menstrual cycle affects objective and subject training parameters, it might be feasible to adjust the training program based on the phase of the menstrual cycle.
Does the menstrual cycle affect recovery? | 2 years
  Improving endurance, muscle strength and power is not only training, but also the quality of recovery. Therefore, it is interesting to investigate whether the hormonal changes during the menstrual cycle affect recovery (i.e. readiness).

OTHER OUTCOMES:
Questionnaires | 3 years
  Out of the complete cohort included, it is possible to select a specific group of cyclist to dive deeper into menstrual cycle related training parameters
Excercise testing | 3 years
  Out of the complete cohort included, it is possible to select a specific group of cyclist who can be invited to perform excercise tests during different moments of the menstrual cycle.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Martini Ziekenhuis, Groningen
  - Martini ziekenhuis, Groningen

IPD SHARING:
Plan to Share IPD: Undecided